CLINICAL TRIAL: NCT06584929
Title: Evaluating Population-Based Strategies for Rural Smoking Cessation
Brief Title: Rural Smoking Cessation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024LS139
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Condition (Experimental): Weekly text and email messages referring to Smokefree.gov, NRT Starter kit, free 2-week supply of patches (Nicoderm CQ in either 21 or 14 mg nicotine) and lozenges (Nicorette Nicotine Lozenges, Mint Flavor in either 4 or 2 mg nicotine) with NRT education plus referral to where to request more NRT.
  Interventions: Drug: Nicoderm CQ nicotine patch; Drug: Nicorette Nicotine Lozenges
- Control Condition (No Intervention): Weekly text and email messages referring to Smokefree.gov
- RHE - Intervention Condition (No Intervention): Weekly text and email messages on reduced harm or exposure (RHE) tobacco products.

INTERVENTIONS:
Drug: Nicoderm CQ nicotine patch — Two week supply provided to participants on study.
  Arms: Intervention Condition
Drug: Nicorette Nicotine Lozenges — Two week supply provided to participants on study.
  Arms: Intervention Condition

SUMMARY:
Understanding ways to help people who live in rural areas quit smoking is a public health priority. quitting smoking among rural people who smoke is a critical public health concern. People in rural areas smoke at higher rates than those in urban areas, experience high rates of smoking caused cancers and deaths. We are recruiting rural people from around the country to better understand how different quit smoking methods can improve a person's chances of successfully quitting smoking.

DETAILED DESCRIPTION:
This is a SMART, where eligible rural people who smoke (RPWS) can be randomized up to two times to different resources/ways to help quit smoking. For each randomization, participants will use the assigned resources for 3 months, and partake in surveys at baseline, 1, and 3 months, during which they will be asked several questions related to use of resources, and smoking behavior. Carbon monoxide (CO) in exhaled breath will be collected at 3 months using iCO™ Smokerlyzer® (https://www.icoquit.com/us/) to determine biochemically confirmed abstinence.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 years
* smoke ≥ 5 cigarettes per day
* daily access to their own iPhone/Android smartphone or tablet

Exclusion Criteria:

* past 30-day NRT use or contraindications listed on the NRT labels
* currently pregnant/breastfeeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants abstinent from all combustible tobacco products | 3 months
  Biochemically-confirmed 7-day abstinence from all combustible tobacco products at 3 months.

SECONDARY OUTCOMES:
Cigarettes per day (CPD) | 1 and 3 months
  Number of cigarettes smoked per day.